CLINICAL TRIAL: NCT03870308
Title: fMRI of Active DBS Stimulation in Epilepsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Erik H. Middlebrooks, M.D., Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18-010321
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Epilepsy
Keywords: Deep Brain Stimulation
MeSH Terms: conditions — Epilepsy | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Deep Brain Stimulation subjects (Experimental)
  Interventions: Diagnostic Test: Functional MRI

INTERVENTIONS:
Diagnostic Test: Functional MRI — A special type of MRI measuring the metabolic changes that occur within the brain. It may be used to examine the brain's anatomy and determine which parts of the brain are handling critical functions. It helps identify important language and movement control areas in the brain.

SUMMARY:
Researchers are trying to incorporate a process known as Functional MRI (fMRI) scanning to reveal a pattern in brain activity during Deep Brain Stimulation (DBS), which will correlate to possible seizure freedom.

ELIGIBILITY:
Inclusion Criteria

* Patients selected to undergo anterior thalamic nucleus DBS for refractory epilepsy

Exclusion Criteria

* Contraindication to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-03-05 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-11 (Actual)

PRIMARY OUTCOMES:
DBS Stimulation | One year
  The primary endpoint of this feasibility study is detection of functional MRI activation related to DBS stimulation.

CONTACTS AND LOCATIONS:
Overall Officials: Erik H Middlebrooks, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials